CLINICAL TRIAL: NCT05488652
Title: Cerebromicrovascular Effects of Time-Restricted Eating in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14856
Record Dates: First submitted 2022-07-22; First posted 2022-08-04 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Time Restricted Eating
Keywords: Time restricted eating; Intermittent fasting; neurovascular coupling; cognitive function; aging
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): no intervention
- Time restricted eating (Experimental): not more than 10 hrs. eating window daily goal for 6 months
  Interventions: Other: Time restricted eating

INTERVENTIONS:
Other: Time restricted eating — not more than 10 hrs. eating window daily goal for 6 months
  Arms: Time restricted eating

SUMMARY:
The central hypothesis of this study is that closer adherence to time restricted eating (TRE) will improve endothelial function, neurovascular (NVC) responses, resulting in improved cognitive performance, potentially through activation of SIRT1-dependent vasoprotective pathways.

DETAILED DESCRIPTION:
This hypothesis will be tested by assessing the effect of TRE (not more than 10hr eating window each day for 6 months) in healthy adults (≥21 years of age). The group of subjects enrolled into TRE arm will be compared to control group. All participants will be randomized into either arm of the study.

ELIGIBILITY:
Inclusion Criteria:

-Healthy adults ≥21 years of age

Exclusion Criteria:

-Inability to read or write in English

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Change in neurovascular coupling using functional near infrared spectroscopy (fNIRS) | baseline, up to 6 months
  Functional near infrared spectroscopy (fNIRS) will be performed during the cognitive n-back task. fNIRS approach generates data that represent a relative change in oxygenated and deoxygenated hemoglobin measured over the cortical brain tissues. Neurovascular coupling will be evaluated as a change in oxy- and deoxy-hemoglobin between before and after treatment.
Change in neurovascular coupling using transcranial Doppler | baseline, up to 6 months
  Transcranial Doppler sonography will be used to measure the change in the blood flow velocities during the cognitive n-back task between before and after treatment.
Change in neurovascular coupling using the dynamic retinal vessel analysis | baseline, up to 6 months
  Flicker light-induced dilation of the retinal vessels (percentage increase over baseline diameter) will be measured in the right or left eye of each study participant using the Dynamic Vessel Analyzer (DVA, IMEDOS Systems, Jena, Germany). The change in retinal vessel diameters is tracked and reported as a %change from baseline, before and after treatment. .

SECONDARY OUTCOMES:
Change in microvascular endothelial function | baseline, up to 6 months
  Changes in microvascular endothelial function will be assessed using laser speckle contrast imaging (LSCI) in the hand using the flow mediated dilation approach. The change in skin perfusion is calculated and reported as a %change from baseline, between before and after treatment.
Change in macrovascular endothelial function | baseline, up to 6 months
  Changes in macrovascular endothelial function will be assessed using sonography during flow mediated dilation approach. The change in brachial artery diameter is calculated and reported as a %change from baseline, between before and after treatment.
Change in deep tissue oxygen saturation | baseline, up to 6 months
  Transcutaneous deep tissue oxygen saturation will be measured using the inSpectra near infrared device. The data are calculated and reported as a %change from baseline, between before and after treatment.
Change in arterial stiffness | baseline, up to 6 months
  The arterial stiffness will be measured using the pulse wave analysis approach (SphygmoCor, Atcor medical, Itasca IL, or similar). Analysis generated the augmentation index which will be used for comparison before and after treatment.
Change in ECG | baseline, up to 6 months
  ECG will be recorded for heart rate variability analysis. The values of high frequency domain, low frequency domain, their ratio, as well as total power will be calculated and used for comparison before and after treatment. .
Change in Glycocalyx - perfused boundary region | baseline, up to 6 months
  Video recordings of the sublingual vasculature will be performed using the high definition video camera GlycoCheck (Microvascular health solutions). Data collected will include perfused boundary region (um), and will be used for comparison before and after treatment.
Change in capillary density | baseline, up to 6 months
  Video recordings of the sublingual vasculature will be performed using the high definition video camera GlycoCheck (Microvascular health solutions). Data collected will include capillary density (mm/mm^2), and will be used for comparison before and after treatment.
Change in red blood cell velocity | baseline, up to 6 months
  Video recordings of the sublingual vasculature will be performed using the high definition video camera GlycoCheck (Microvascular health solutions). Data collected will include red blood cell velocity (um/sec), and will be used for comparison before and after treatment.
Change in Attention | baseline, up to 6 months
  The allocation of one's limited capacities to deal with an abundance of environmental stimulation will be measured in a combined "Flanker Inhibitory Control and Attention Test".Units of measure - score (from 0 to 10, bigger number is better). Reported as a %change from baseline, before and after treatment.
Change in Episodic Memory | baseline, up to 6 months
  Cognitive processes involved in the acquisition, storage and retrieval of new information, will be measured using the "Picture Sequence Memory Test". Unit of measure - overall score (bigger number is better). Reported as a %change from baseline, before and after treatment.
Change in Working Memory | baseline, up to 6 months
  The ability to store information until the amount of information to be stored exceeds one's capacity to hold that information will be measured using the "List Sorting Working Memory Test". Unit of measure - overall score (bigger number is better). Reported as a %change from baseline, before and after treatment.
Change in Language | baseline, up to 6 months
  Picture Vocabulary Test measures receptive vocabulary administered in a computer-adaptive test (CAT) format. Respondents select the picture that most closely matches the meaning of the word, before and after treatment. Unit of measure - overall score (bigger number is better). Reported as a %change from baseline, before and after treatment.
Change in Executive Function | baseline, up to 6 months
  The capacity to plan, organize and monitor the executive of behaviors that are strategically directed in a goal-oriented manner, will be measured using the "Dimensional Change Card Sort Test". Units of measure - score (from 0 to 10, bigger number is better). Reported as a %change from baseline, before and after treatment.
Change in Processing Speed | baseline, up to 6 months
  Pattern Comparison Processing Speed Test assesses the amount of information that can be processed within a certain unit of time. Items are simple so as to purely measure processing speed. Units of measure - score (from 0 to 130, bigger number is better). Reported as a %change from baseline, before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Tarantini, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No